CLINICAL TRIAL: NCT04973150
Title: Study on the Effect of Eye-covering Pretreatment on Acute Delirium After General Anesthesia in Pre-school Aged Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, DONG Peifang, Head nurse, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: dpf199438
Record Dates: First submitted 2021-06-20; First posted 2021-07-22 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Ophthalmology
Keywords: Pre-school Aged Children; Acute Delirium; Eye-covering Pretreatment
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the children were given gauze covering training in one eye or both eyes (Experimental): According to the operation method, the children were given gauze covering training in one eye or both eyes.
  Interventions: Behavioral: To explore whether pretreatment with eye covering can reduce the incidence of acute delirium and the score of delirium after general anesthesia in ophthalmology pre-age children.
- Using regular tablet computer to play cartoon animation video (No Intervention)

INTERVENTIONS:
Behavioral: To explore whether pretreatment with eye covering can reduce the incidence of acute delirium and the score of delirium after general anesthesia in ophthalmology pre-age children. — To explore whether pretreatment with eye covering can reduce the incidence of acute delirium and the score of delirium after general anesthesia in ophthalmology pre-age children. Methods A total of 300 preschool-age children who underwent general anesthesia of selective ophthalmic surgery in a 3A grade hospital from August 2019 to July 2020 were selected as the research object, who were divided into experimental group and control group with 150 cases each by random number table. Children in the control group received regular education on cartoon animation videos before surgery; children in the experimental group received eye-covering pretreatment on the basis of cartoon animation videos. The differences in preoperative anxiety degree score, postoperative acute delirium incidence, delirium degree score, and postoperative nursing care difficulty score were compared between the two groups.
  Arms: the children were given gauze covering training in one eye or both eyes

SUMMARY:
Participants (preschool children), because their cognitive ability and anti pressure ability are obviously weaker than adults, most of the children who have this kind of operation and anesthesia stressors will have perioperative anxiety. After eye surgery, they need to bandage their eyes with gauze (single or double), so that the participants are in a state of complete or partial darkness for a certain period of time, which is easy to produce dark phobia. In clinical practice, investigators found that more than 80% of children with advanced ophthalmology were prone to leprosy, resistance, crying and other symptoms after general anesthesia, which brought greater difficulties to nursing. How to improve the cognitive ability of preschool children, reduce the anxiety level of children during the perioperative period, the incidence of postoperative detention and the difficulty of nursing are new topics worthy of exploration.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 3-7;
2. Selective ophthalmological general anesthesia (static inhalation compound: propofol + fentanil intravenous administration; heptaflurane inhalation);
3. No mental disorders, stunting and low intelligence;
4. There is no other history of surgical hospitalization.

Exclusion Criteria:

1. Those who have completed the operation under local anesthesia;
2. People with visual impairment of both eyes;
3. Eyeball removal and/or eye socket implanter;
4. Hearing and language impairment cannot communicate normally;
5. Have a history of taking psychotropic drugs;
6. People with severe organs such as the heart, lungs, brains and kidneys.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 350 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety | Up to 24 weeks
  The modified Yale preoperative anxiety scale (m-ypas) was used to evaluate the preoperative anxiety. The scale has high reliability and validity (Cronbach's) α The reliability coefficient was 0.936; 91). The scale is often used to evaluate the preoperative anxiety level of children aged 2-12 in the waiting room, going to the operating room, entering the operating room and anesthesia induction period. The questionnaire consists of 5 parts and 22 items, which are language (4 items), vocalization (6 items), emotional expression (4 items), obvious alertness (4 items), and the role of parents (4 items). In addition to the vocal part of 1-6 points, the rest are 1-4 points, the minimum is 0 points, the maximum is 100 points, the higher the score, the higher the anxiety level of the subjects. The scale was evaluated by the anesthesiologist when the child entered the operating room, and the evaluation time was about 2 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- peifang Dong, Hangzhou, China

REFERENCES:
- [Derived] Dong PF, Qiao DN, Chen HL, Lu SH, Qu SH, Wu YT, Zhao D, Wan T. Effect of Different Durations of Eye-Covering Pretreatment on Emergence Delirium after Ophthalmic Surgery in Preschool-Aged Children: A Randomized Controlled Study. J Ophthalmol. 2022 Sep 16;2022:3656148. doi: 10.1155/2022/3656148. eCollection 2022. PMID 36157681